CLINICAL TRIAL: NCT06688006
Title: The Effect of Climate Change Education and a Short Animated Film on Pregnant Women's Awareness and Hope Levels: A Randomized Controlled Trial
Brief Title: Climate Change Education and a Short Animated Film on Pregnant Women's Awareness and Hope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Yasemin ERKAL AKSOY, Assoc. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 29051453
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Awareness; Pregnancy Related; Hope
Keywords: climate change; short animated film

STUDY DESIGN:
Intervention Model Description: To ensure randomization in the study, the blocks will first be created by stratifying the pregnant women according to their age and level of education using the stratified sampling method, and then it will be decided whether the pregnant women in the groups will be in the intervention or control group using simple randomization. Then, a table of random numbers between 1-288 will be generated using the Random.org website with simple random sampling method (https://www.random.org/sequences/).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The generated numbers are written on small pieces of paper, folded and placed in a small box. The box will be given to the pregnant woman by a midwife not involved in the study and she will be asked to draw a number. This will determine whether the pregnant woman is in the intervention group or the control group. This reduces the possibility of bias in the study. During the data collection process of the study, the researcher will know which group the pregnant women are in, but the pregnant women will not know which group they are in. A single-blind method will be used. The statistics of the trial will be done by a statistician who is not involved in the trial. The intervention and control groups will be given a code or colour so that the statistician does not know which group the data belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: climate change short animation film (Experimental): Before enrolling the pregnant women in the intervention group, the informed consent form, the personal information form, the climate change awareness scale for pregnant women and the climate change hope scale (pre-test) will be completed. The researcher will then give a 30-minute training presentation on the climate crisis to the pregnant women individually in the conference room on the third floor of the maternity hospital. Two weeks after the training, the worker will open a meeting session via Microsoft Teams or Google Meet, and a short animated film will be watched on this platform as a reminder. Four weeks after the viewing of the short animation film, another meeting session will be set up via Microsoft Teams or Google Meet and the link to the survey form will be shared online and the final evaluations (post-test - questions on climate change, climate change awareness scale and hope scale for preventing climate change) will be carried out.
  Interventions: Other: climate change short animation film
- Control (No Intervention): No application will be made to the pregnant women in the control group, and the informed consent form, personal information form, Climate Change Pregnancy Awareness Scale and Climate Change Prevention Hope Scale (pre-test) will be completed at the first interview. During this time, a sign will be hung on the door to prevent anyone from entering or leaving the room. Six weeks after the first interview, the link to the survey form (Questions about Climate Change, Climate Change Pregnant Awareness Scale and Climate Change Prevention Hope Scale) will be shared with the pregnant women via Microsoft Teams or Google Meet and their final evaluation (post-test) will be conducted. A video interview will be conducted with the control group in a Microsoft Teams or Google Meet meeting to ensure that real people completed the form. At the end of the study, an educational booklet and a short animated film on climate change will be sent online.

INTERVENTIONS:
Other: climate change short animation film — For the short animated film, a scenario will be created that describes climate change, risk factors that threaten human health as a result of climate change, adverse health effects of climate change, adverse effects on maternal and foetal health, precautions to be taken to protect against and adapt to the adverse effects of climate change. In the short animation film, visual materials will be created that show the adverse effects of climate change by using developing technology. The created scenario will be prepared as a two-dimensional (2D) animation film with the support of Selçuk University SERATEM (Selçuk University Radio and Television Application Center). All lines, colours, decorations and characters used in the creation phase of the short animation film will be determined by the researchers. Once the drawing and animation phases are complete, the voice-over actors will be selected after a further review. The short animated film should be about 2-3 minutes long.
  Arms: Experimental: climate change short animation film

SUMMARY:
Pregnant women are among the groups most affected by the negative health effects of climate change, such as low birth weight, preterm birth, premature rupture of membranes, stillbirth, gestational diabetes, gestational hypertension and preeclampsia, spontaneous abortion, malnutrition, respiratory illness and stress, depression, post-traumatic stress disorder. It can lead to adverse pregnancy outcomes, including psychological problems. Climate change education enables pregnant women to make informed decisions by raising their awareness and helps improve their ability to adapt to the negative effects of climate change. Health education for individuals and pregnant women uses methods such as demonstration, role-playing, screening, expression, question-answering, problem-solving, and short animated films. Short animated films, which are visual and auditory media and are an interesting method of health education, ensure that the information conveyed is stored in long-term memory. No studies were found in Turkey to determine pregnant women's awareness and hope regarding climate change or to increase their awareness and knowledge through education and short animated films. The creation of an original short animated film and its support through education show the difference of this study from other studies. Therefore, this study was planned based on the assumption that climate change education and short animated film would increase the awareness and hope of pregnant women. The purpose of this study is to investigate the effects of climate change education and short animated film on pregnant women's awareness and hope. This study was designed as a randomized controlled trial.

DETAILED DESCRIPTION:
The population of the study is all pregnant women in the second and third trimesters who present to the antenatal clinic of Konya City Hospital. The sample of the study consists of pregnant women who meet the criteria for inclusion in the study and agree to participate in the study after being informed about the study. G-Power 3.1.9.7, based on the Hope Scale for the Prevention of Climate Change score average (56.14±9.75), of which the study sample size is known. The program calculated the 3-unit difference by choosing a power of 0.85, an effect size of 0.30, an alpha level of 0.05, and a two-sided hypothesis option, and aimed to reach a total of 262 participants, 131 in the intervention group and 131 in the control group. Considering the data loss, it was planned to conduct the study with 276 pregnant women, which is 5% more than the set sample number. Research data: collected on a self-report basis using the "Informed Consent Form"," the "Personal Information Form"," the "Pregnant Awareness Scale for the Effects of Climate Change on Maternal Fetal Health," and the "Climate Change Hope Scale"." Pre-tests with questionnaires will be conducted at the first interview with the pregnant women who were randomly assigned to the intervention and control groups. An educational brochure on climate change will be given to the pregnant women in the intervention group, and a presentation will be given by the researcher. Two weeks after the training, a short animated film will be viewed via WhatsApp as a reminder. Two weeks after watching the short animated film, the link to the survey form will be shared online via WhatsApp, and final evaluations will be conducted. Pregnant women who are part of the control group will not undergo any intervention application. Four weeks after the first meeting, a link to the survey form will be shared via WhatsApp and final evaluations will be conducted. After completion of the study, the educational brochure and the short animated film on climate change will be sent online to the pregnant women in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-49,
* Have a singleton pregnancy,
* Have at least a primary school education and are able to communicate,
* Have no vision or hearing problems
* and use an online communication platform (Microsoft Teams or Google Meet)

Exclusion Criteria:

* Pregnant women who conceived with assisted reproductive techniques and have high-risk pregnancies
* Pregnant women who received training during the study but did not watch the short animated film on Microsoft Teams and Google Meet,
* who gave birth,
* who wanted to leave

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 288 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Personality Information Form | Baseline (at the beginning of the study)
  The personal information form is a questionnaire developed by the researchers based on the literature. The survey includes 13 questions on the introductory socio-demographic characteristics (age, education, etc.) of women and their husbands, 16 questions on the obstetric characteristics of women (gestational week, number of pregnancies, etc.), and 18 questions on climate change (Ha et al. 2018, Kısrık and Avcıbay Vurgeç 2022, Leung et al. 2023).
Climate Change Pregnant Awareness Scale | Baseline (at the beginning of the study)
  The Climate Change Pregnant Awareness Scale is a 21-item scale developed by Kısrık and Avcıbay Vurgeç (2022) to assess pregnant women's awareness of the effects of climate change on maternal-fetal health. Each of the scale items is a 5-point Likert-type item as "1-I strongly disagree, 2-I partially disagree, 3-I am undecided, 4-I slightly agree, 5-I strongly agree". There is no reverse item in the scale. It consists of 3 subscales: General (items 1, 2, 3, 4, 7 and 8), Fetal (items 5, 6, 11, 12, 13, 14 and 15 and 16) and Maternal (items 9, 10, 17, 18, 19, 20 and 21). The score obtained for each sub-dimension indicates awareness of that sub-dimension. The minimum score for the total scale is 21 and the maximum is 105. As the total score increases, women's awareness of climate change increases. The overall Cronbach's alpha coefficient of the scale is 0.94.
Climate Change Pregnant Awareness Scale | six weeks after education
  The Climate Change Pregnant Awareness Scale is a 21-item scale developed by Kısrık and Avcıbay Vurgeç (2022) to assess pregnant women's awareness of the effects of climate change on maternal-fetal health. Each of the scale items is a 5-point Likert-type item as "1-I strongly disagree, 2-I partially disagree, 3-I am undecided, 4-I slightly agree, 5-I strongly agree". There is no reverse item in the scale. It consists of 3 subscales: General (items 1, 2, 3, 4, 7 and 8), Fetal (items 5, 6, 11, 12, 13, 14 and 15 and 16) and Maternal (items 9, 10, 17, 18, 19, 20 and 21). The score obtained for each sub-dimension indicates awareness of that sub-dimension. The minimum score for the total scale is 21 and the maximum is 105. As the total score increases, women's awareness of climate change increases. The overall Cronbach's alpha coefficient of the scale is 0.94.

SECONDARY OUTCOMES:
Hope for Preventing Climate Change Scale (HOC) | Baseline (at the beginning of the study)
  In a global crisis such as climate change, individuals' hopes can increase their active participation in finding solutions to mitigate and adapt to climate change (Sangervo et al. 2022). The Hope for Prevention of Climate Change Scale (HOC) was developed by Li and Monreo (2018) to measure individuals' hope for preventing and combating climate change (Li and Monreo 2018). Li and Monreo (2018); emphasise that the scale can be used by researchers who want to use a quantitative approach to investigate climate change hopes, or to test the effectiveness of climate change education programmes to increase individuals' climate action. The use of the scale is particularly important in awareness-raising and education programmes in terms of measuring not only individuals' knowledge about climate change, but also their motivation and belief that they can turn this knowledge into action (Li and Monroe 2018).
Hope for Preventing Climate Change Scale (HOC) | six weeks after education
  In a global crisis such as climate change, individuals' hopes can increase their active participation in finding solutions to mitigate and adapt to climate change (Sangervo et al. 2022). The Hope for Prevention of Climate Change Scale (HOC) was developed by Li and Monreo (2018) to measure individuals' hope for preventing and combating climate change (Li and Monreo 2018). Li and Monreo (2018); emphasise that the scale can be used by researchers who want to use a quantitative approach to investigate climate change hopes, or to test the effectiveness of climate change education programmes to increase individuals' climate action. The use of the scale is particularly important in awareness-raising and education programmes in terms of measuring not only individuals' knowledge about climate change, but also their motivation and belief that they can turn this knowledge into action (Li and Monroe 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No